CLINICAL TRIAL: NCT01345916
Title: A Phase 3,8-week Clinical Trial to Test the Efficacy of CHF1535 Via NEXT DPI® Versus Same Dose of CHF1535 pMDI and Beclomethasone DPI 100µg on PEF in Adult Asthmatic Patients After 1 Month of Treatment With FOSTER®
Brief Title: Efficacy of CHF1535 Via NEXT DPI Versus pMDI and BDP DPI100µg on PeakExpiratoryFlow in Asthmatic Patients
Acronym: Neptune
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCD-1009-PR-0050; 2010-023281-47 (EudraCT Number)
Record Dates: First submitted 2011-04-12; First posted 2011-05-02 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHF 1535 100/6 NEXT Dry Powder Inhaler® (Experimental): CHF1535 100/6 NEXT DPI® 1 inhalation bis in day (b.i.d) (daily dose BDP 200/FF 12 µg)
  Interventions: Drug: CHF 1535 100/6 NEXT DPI® 2 months
- CHF1535 100/6 pMDI (Active Comparator): CHF1535 100/6 pressurisedMeterDoseInhaler 1 inhalation b.i.d (total daily dose BDP 200/FF 12 µg)
  Interventions: Drug: CHF 1535 100/6 pMDI 2 months
- beclomethasone dipropionate DPI (Active Comparator): beclomethasone dipropionate 100 µg DPI, 1 inhalation b.i.d (total daily dose BDP 200 µg)
  Interventions: Drug: BDP DPI 2 months

INTERVENTIONS:
Drug: CHF 1535 100/6 NEXT DPI® 2 months — CHF 1535 100/6 NEXT DPI® 2 months
  Arms: CHF 1535 100/6 NEXT Dry Powder Inhaler®
Drug: CHF 1535 100/6 pMDI 2 months — CHF 1535 100/6 pMDI 2 months
  Other Names: Foster®
  Arms: CHF1535 100/6 pMDI
Drug: BDP DPI 2 months — BDP DPI 2 months
  Other Names: Clenil® Pulvinal®
  Arms: beclomethasone dipropionate DPI

SUMMARY:
The purpose of this study is to demonstrate that CHF 1535 NEXT DPI® is non-inferior to the corresponding dose of CHF 1535 pMDI and superior to marketed beclomethasone DPI 100 µg in terms of average pre-dose morning Peak Expiratory Flow (PEF) in asthmatic adult patients.

DETAILED DESCRIPTION:
The primary objective is to demonstrate that CHF 1535 NEXT DPI® (beclomethasone dipropionate + formoterol fumarate 100/6 μg), 1 inhalation twice daily, is non-inferior to the corresponding dose of CHF 1535 pMDI in terms of pulmonary function test (change from baseline to the entire treatment period in average pre-dose morning PEF) in asthmatic adult patients ≥ 18 years under treatment with fixed dose combination of Foster® (beclomethasone dipropionate + formoterol fumarate 100 / 6 μg) 1 inhalation bid.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults (≥18 years old).
2. Reversibility test defined as ΔFEV1 ≥ 12% and ≥ 200 mL .
3. FEV1 > 80% of the predicted values .
4. Asthma Control Questionnaire score < 1.25.
5. Asthmatic patients
6. Non- or ex-smokers

Exclusion Criteria:

1. History of near fatal asthma.
2. COPD patients
3. Asthma exacerbation within 1 month prior to the screening visit or asthma exacerbation during the run-in period.
4. Lower respiratory tract infection within 1 month prior Visit1 (V1).
5. History of cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency.
6. Diagnosis of restrictive lung disease.
7. Patients treated with oral or parenteral corticosteroids in the previous 2 months before V1
8. Intolerance or contra-indication to treatment with beta 2-agonists and/or inhaled corticosteroids or allergy to any component of the study treatments.
9. Significant medical history of and/or treatments
10. Active cancer or a history of cancer .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 932 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the entire treatment period in average pre-dose morning Peak Expiratory Flow. | at 8 weeks

SECONDARY OUTCOMES:
Pre-dose morning FEV1 (Forced Expiratory Volume in one second); | at 2, 4, 6 and 8 weeks of treatment
Pre-dose morning FVC (Force Vital Capacity) ; | at 2, 4, 6 and 8 weeks of treatment
ACQ (Asthma Control Questionnaire) score ; | at eight weeks
pre-dose evening PEF ; | at 2, 4, 6 and 8 weeks of treatment
daily PEF variability ; | at 2, 4, 6 and 8 weeks of treatment
use of rescue medication ; | at 2, 4, 6 and 8 weeks of treatment
percentage of rescue use-free days | at 2, 4, 6 and 8 weeks of treatment
pre-dose morning PEF ; | at 2, 4, 6 and 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frank KANNIESS, Dr, Principal Investigator — Gemeinschaftspraxis Reinfeld - Raiffeisenpassage 15 - D-23858 Reinfeld - Germany
Locations (1):
- GSPZOZ Uniwersytecki Szpital Kliniczny, Lodz, Poland

REFERENCES:
- [Result] Kanniess F, Scuri M, Vezzoli S, Francisco C, Petruzzelli S. Extrafine beclomethasone/formoterol combination via a dry powder inhaler (NEXThaler((R))) or pMDI and beclomethasone monotherapy for maintenance of asthma control in adult patients: A randomised, double-blind trial. Pulm Pharmacol Ther. 2015 Feb;30:121-7. doi: 10.1016/j.pupt.2014.07.006. Epub 2014 Aug 1. PMID 25088067
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-023281-47